CLINICAL TRIAL: NCT04453475
Title: Therapies to Achieve Treatment Goals While Being Exposed to Hygiene and Distance Rules: Feasibility and Benefits of Digital Services During the COVID19 Pandemic (Anhand-COVID19)
Brief Title: Feasibility and Benefits of Digital Services During the COVID19 Pandemic
Acronym: AnhandCOV19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: Dr. Becker Hospital Group (Other); Dr. Becker Burg-Klinik (Burg) (Unknown); Dr. Becker Klinik Norddeich (NOR) (Unknown); Dr. Becker Klinik Juliana (JUL) (Unknown); Dr. Becker Klinik Möhnesee (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Anhand-COVID19
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Psychosomatic Disorder; Psychological Distress; Psychological Stress; Psychological Disease; Psychological Disorder; Psychological Impairment; Psychological Disability; Psychological Adjustment; Psychological Adaptation; Communication; Health Care Seeking Behavior; Anxiety; Behavior, Health; Health Risk Behaviors; Healthy Lifestyle
Keywords: health behavior change; stress; eHealth; digital intervention; medical rehabilitation; clinic stay
MeSH Terms: conditions — Psychophysiologic Disorders; Stress, Psychological; Mental Disorders; Communication; Patient Acceptance of Health Care; Anxiety Disorders; Health Behavior; Health Risk Behaviors | interventions — Health Literacy

STUDY DESIGN:
Intervention Model Description: The methodology uses a natural variation design within the Dr. Becker Clinical Group. The interventions consist of an online depression session as a "flipped classroom" and/or an online lecture with socio-medical content, which are combined in such a way that the differential effects can be evaluated. For this purpose, a control group is included that does not receive these two interventions (but receives a similar rehabilitation treatment to the intervention groups).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Partial digital group: depression (Experimental): Burg
  Online depression session as a "flipped classroom" and voluntary low-threshold communication trainings as well as training on rehabilitation goals
  Interventions: Behavioral: Training session adressing information and health literacy
- Partial digital group: social work (social medicine) (Experimental): NOR
  Online lecture with socio-medical content and voluntary low-threshold communication trainings as well as training on rehabilitation goals
  Interventions: Behavioral: Training session adressing information and health literacy
- Partial digital group: depression + social work (Experimental): JUL
  Online depression session as a "flipped classroom" and an online lecture with socio-medical content and voluntary low-threshold communication trainings as well as training on rehabilitation goals
  Interventions: Behavioral: Training session adressing information and health literacy
- Control group: only digital training before rehabilitation (Active Comparator): MOE
  Online tobacco cessation a "flipped classroom" and voluntary low-threshold communication trainings as well as training on rehabilitation goals
  Interventions: Behavioral: Training session adressing information and health literacy

INTERVENTIONS:
Behavioral: Training session adressing information and health literacy — The training sessions are provided online and as alternative to face-to-face treatments which cannot be provided as before due to the safety regulations relating to Covid-19

SUMMARY:
As a result of the pandemic, hygiene and distancing rules must be followed in Health care/ rehabilitation clinics to ensure the safety of patients and staff. This has led to extensive changes in the therapy processes, including a reduction in group sizes and maintaining distances within the groups, resulting in a reduction in the range of therapies available to individuals, since the number of employees remains unchanged and cannot be increased at will and in the short term due to the lack of qualified staff. In order for the treatment/rehabilitation goals to be achieved nonetheless, new forms of implementation of therapy programs must be developed in addition to organizational adjustments. Digitalization can be a significant support in this respect. The majority of patients in psychosomatic rehabilitation possess smartphones, meaning that the necessary infrastructure for the utilization of digital offers is available and can be used to the greatest possible extent. The use of digital measures within the therapeutic services supports the independence of the patients, as they can use the digital offers independently and flexibly in their own time.

How should Health care/rehabilitation services be designed in light of the SARS-CoV-2 pandemic and which services have the potential to buffer future crises: What general recommendations can be derived for the design of such services for routine care? What are support measures to encourage social participation and return to work?

DETAILED DESCRIPTION:
In Germany, the SARS-CoV-2 pandemic represents a crisis with massive effects on health and rehabilitation care. This crisis is not a short-term event but will also has longer-term effects on health care service/rehabilitation. Necessary adjustments due to hygiene and distance regulations include, for example, the reduction of group sizes and alternatives to conventional service provision (= digital services, McNeary et al., 2020). How such offers are perceived and accepted by patients and staff is crucial for the effect on the care. Systematic research into the pandemic from the patient and employee perspective, its consequences for procedures in rehabilitation clinics and for the implementation of the necessary therapies is required in a timely manner in order to better understand and mitigate the effects of the pandemic and to ensure the effectiveness of rehabilitation. This is the aim of this project with a focus on digital services and their subjective usefulness.

Furthermore, the integration of such offers can mean that a therapist is not present during the entire therapy, but that rehabilitants first learn the basics of a topic in self-study. This is based on the principle of the "Flipped Classroom". (Rehab) Patients as well as employees of the clinics are involved in the piloting of the survey instruments and the final choice of outcome criteria as well as the derivation of possible applications (guidelines, recommendations for rehabilitants).

In addition, the pandemic is negatively associated with equal participation of vulnerable groups (e.g. persons with physical or psychological handicaps). In the case of medical rehabilitation patients, particular occupational problems make equal participation and social cohesion more difficult: problems such as long-term limited productivity or the threat of exclusion from the labor market (pension for reduced earning capacity), negative employment forecasts and experiences of previously limited social participation are in turn further exacerbated by demographic change and the consequences of the COVID 19 pandemic. These restrictions are also reflected in the increased experience of loneliness. To date, however, there is a lack of a systematic understanding of these circular, dynamic processes and low-threshold, effective approaches to action, effective approaches to action.

The following questions will be empirically investigated:

1. How are digital services evaluated regarding feasibility, acceptance and subjective usefulness in light of the current situation?
2. Which characteristics of rehabilitants are related to the acceptance and subjective usefulness of digital offers?
3. For which patients of rehabilitation is there a need for support in the use of digital services to achieve rehabilitation goals?
4. Are there differences in perceived usefulness between services?
5. How do people in the welfare state and labor market with disabilities and impairments (rehabilitants) perceive the consequences of the Covid 19 pandemic and the transformation processes?
6. How effective are support measures with regard to communication for rehabilitants in supporting equal participation?
7. How should support for equal participation be designed in the long term: What What are the consequences for labor market and social policy?

The methodology uses a natural variation design within the Dr. Becker Clinical Group in order to investigate the issues at the highest possible scientific level and to achieve reliable results. The interventions consist of an online depression session as a "flipped classroom" and/or an online lecture with socio-medical content, and/ or a tobacco cessation lecture, which are combined in such a way that the differential effects can be evaluated. For this purpose, a control group is included that does not participate in these interventions (but receives the standard rehabilitation treatment programm). Furthermore, all groups voluntarily receive patient training before rehabilitation with the content of setting "treatment goals" as well as an invitation to pre- and post-surveys.

The survey methods are online surveys (before the treatment=pre (T1); end of treatment=post (T2); end of treatment=post 12 weeks (T3)) by means of UniPark.

The main target variables are reported behavior and well-being (stress/burden of COVID-19 disease or probability of disease, limitations, quality of life, anxiety or depression; pre-post comparison) as well as subjective need (pre) and benefit (post) of the digital services. Further primary target variables are concentrated on social participation, workability and return to work. The theoretical foundation for the selection of target variables and constructs is the Carry-Over Action Model. The sample includes all rehabilitands who undergo a psychosomatic rehabilitation in the hospitals. The planned sample size of the rehabilitants is N = 2,000.

The feasibility is given by the use of an existing care system with cover letters from the patients before the treatment. Possible disturbance variables such as affinity towards technology (which could lead to a lower participation rate among participants with little affinity towards technology) are controlled for and taken into account in the evaluation. Gender and diversity are considered as covariates or moderators in the statistical models.

All data of the participants will be treated in accordance with the data security regulations (DSGVO), good scientific practice and the ethical requirements. Furthermore, all patients are informed about the project, ethics and data protection in a generally understandable way by a cover letter from their clinic before the treatment. All project staff are obliged to comply with the ethics guidelines and to maintain confidentiality. The pre- and post-data of the patients are combined by means of a personal code, which does not allow any conclusion about the participant.

The results of this study will show which digital implementation forms of therapy offers are feasible in terms of benefit and acceptance and can thus contribute to the further development of health care services and medical rehabilitation. This will create the necessary evidence base to include digital offers in the classification of therapeutic services and the therapy standards based on them and thus to establish them in routine care. Furthermore, a guideline for the future integration of these services into the health care services/rehabilitation process will be developed. Due to the standardized combination of analogue and digital therapy parts, therapy goals can be achieved more efficiently on the basis of the validated pedagogical concepts used and with the involvement of fewer human resources. This is not only relevant during the SARS-CoV-2 pandemic, but also with regard to the relevant shortage of qualified personnel. Furthermore, the research basis for digital measures to support social support for social participation will be created. With these findings, similar measures on other groups, for example, persons with disabilities or limitations, can be researched.

ELIGIBILITY:
Inclusion Criteria:

* Patients before the start of the treatment
* Selected by the clinic
* Invited to participate in the study

Exclusion Criteria:

* Inability to read and write
* Severe dementia
* unwillingness to participate in the study and to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Interest in digital interventions (attitudes, behavioral intentions, behavioral experiences) | T1 (prior/beginning of rehab/clinic stay); T2 (end of rehab/clinic stay approx. 5 weeks after T1)
  Quantitative online questionnaire Survey using UniPark
Usability and effectiveness of digital interventions | T1 (prior/beginning of rehab/clinic stay); T2 (end of rehab/clinic stay approx. 5 weeks after T1)
  Quantitative online questionnaire Survey using UniPark
Stressors and barriers due to Covid-19 | T1 (prior/beginning of rehab/clinic stay); T2 (end of rehab/clinic stay approx. 5 weeks after T1)
  Quantitative online questionnaire Survey using UniPark

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Principal Investigator — Jacobs University Bremen
Locations (1):
- Jacobs University Bremen gGmbH, Bremen, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be published. Other researchers are welcome to get in contact with the PI to get access to anonymous data.

REFERENCES:
- [Background] Baumeister, H., Reichler, L., Munzinger, M., & Lin, J. (2014). The impact of guidance on Internet-based mental health interventions - A systematic review. Internet Interventions, 1(4), 205-215. <br /> Direito, A., Carraça, E., Rawstorn, J., Whittaker, R., & Maddison, R. (2017). mHealth technologies to influence physical activity and sedentary behaviors: behavior change zechniques, systematic review and meta-analysis of randomized controlled trials. Annals of Behavioral Medicine, 51, 226-239. doi: 10.1007/s12160-016-9846-0 <br /> Elbert, N. J., Van Os-Medendorp, H., van Renselaar, W., Ekeland, A. G., Hakkaart-van Roijen, L., Raat, H., … Gma, S. (2014). Effectiveness and cost-effectiveness of eHealth interventions in somatic diseases: a systematic review of systematic reviews and meta-analyses. Journal of Medical Internet Research, 16, e110. doi: 10.2196/jmir.2790 <br /> Fleig, L., Lippke, S., Pomp, S., & Schwarzer, R. (2011). Intervention effects of exercise self-regulation on physical exercise and eating fruits and vegetables: a longitudinal study in orthopedic and cardiac rehabilitation. Preventive Medicine, 53, 182-187. <br /> Fleig, L., Pomp, S., Schwarzer, R., & Lippke, S. (2013). Promoting exercise maintenance: How interventions with booster sessions improve long-term rehabilitation outcomes. Rehabilitation Psychology, 58, 323-333. <br /> Granja, C., Janssen, W., & Johansen, M. A. (2018). Factors determining the success and failure of eHealth interventions: systematic review of the literature. Journal of Medical Internet Research, 20, e10235. doi: 10.2196/10235 <br /> Hong, Z., Li, N., Li, D., Li, J., Li, B., Xiong, W., Lu, L., Li, W., & Zhou, D. (2020). Telemedicine during the COVID-19 pandemic: experiences from Western China. Journal of Medical Internet Research, 22, e19577. <br /> Lippke, S., Preißner, C., & Whittal, A. (2018). Facilitating health literacy and behavior change by computer-tailored interventions. In: A. K. Mayer (Ed.). Health Literacy Across the Life (pp. 39-58). Lengerich: Pabst Science Publishers. <br /> Lustria, M. L. A., Noar, S. M., Cortese, J., Van Stee, S. K., Glueckauf, R. L., & Lee, J. (2013). A meta-analysis of web-delivered tailored health behavior change interventions. Journal of Health Communication: International Perspectives, 18, 1039-1069. doi: 10.1080/10810730.2013.768727 <br /> McNeary, L., Maltser, S., Verduzco-Gutierrez, M. (2020). Navigating coronavirus disease 2019 (Covid-19) in physiatry: a CAN report for inpatient rehabilitation facilities. PM R, 12, 512-515. doi:10.1002/pmrj.12369 <br /> Milne-Ives, M., Lam, C., De Cock, C., Van Velthoven, M. H., & Meinert, E. (2020). Mobile apps for health behaviour change in physical activity, diet, drug and alcohol use, and mental health: a systematic review. JMIR Mhealth Uhealth, 8, e17046. doi: 10.2196/17046 <br /> Padala, P. R., Jendro, A. M., & Padala, K. P. (2020). Conducting clinical research during the COVID-19 pandemic: investigator and participant perspectives. JMIR Public Health Surveillance, 6, e18887. <br /> Pérez Sust, P., Solans, O., Fajardo, J.C., Medina Peralta, M., Rodenas, P., Gabaldà, J., Garcia Eroles, L., …, Piera-Jimenez, J. (2020). Turning the crisis into an opportunity: Digital health strategies deployed during the COVID-19 outbreak. JMIR Public Health Surveillance, 6, e19106. <br /> Schuler, M., Murauer, K., Stangl, S., Grau, A., Gabriel, K., Podger, L., . . . Faller, H. (2019). Pre-post changes in main outcomes of medical rehabilitation in Germany: Protocol of a systematic review and meta-analysis of individual participant and aggregated data. BMJ Open, 9. doi:10.1136/bmjopen-2018-023826 <br /> Sheehy, L. M. (2020). Considerations for postacute rehabilitation for survivors of COVID-19. JMIR Public Health Surveillance, 6, e19462. <br /> Storm, V., Dörenkämper, J., Reinwand, D., Wienert, J., De Vries, H., & Lippke, S. (2016). Effectiveness of a web-based computer-tailored multiple-lifestyle intervention for people interested in reducing their cardiovascular risk: A randomized controlled trial. Journal of Medical Internet Research, 18, e78. <br /> Vugts, M. A. P., Joosen, M. C. W., van der Geer, J. E., Zedlitz, A. M. E. E., & Vrijhoef, H. J. M. (2018). The effectiveness of various computer-based interventions for patients with chronic pain or functional somatic syndromes: A systematic review and meta-analysis. PLoS ONE, 13, e0196467. https://doi.org/10.1371/journal.pone.0196467 <br /> Weisel, K. K., Fuhrmann, L. M., Berking, M., Baumeister, H., Cuijpers, P., & Ebert, D. D. (2019). Standalone smartphone apps for mental health - a systematic review and meta-analysis. npj Digital Medicine, 2, 1-10.
- [Result] Keller FM, Dahmen A, Derksen C, Kotting L, Lippke S. Psychosomatic Rehabilitation Patients and the General Population During COVID-19: Online Cross-sectional and Longitudinal Study of Digital Trainings and Rehabilitation Effects. JMIR Ment Health. 2021 Aug 26;8(8):e30610. doi: 10.2196/30610. PMID 34270444
- [Result] Keller FM, Dahmen A, Derksen C, Kotting L, Lippke S. Implementing Digital Trainings within Medical Rehabilitations: Improvement of Mental Health and Synergetic Outcomes with Healthcare Service. Int J Environ Res Public Health. 2021 Aug 25;18(17):8936. doi: 10.3390/ijerph18178936. PMID 34501524
- [Result] Dahmen A, Keller F, Kotting L, Derksen C, Lippke S. [Fear of Coronavirus, Intention to Follow the AHA Rules and Risk Perception Regarding Visits to the Doctor: Cross-sectional Study with Patients suffering from Pre-existing Mental Illness]. Gesundheitswesen. 2021 Apr;83(4):274-281. doi: 10.1055/a-1397-7214. Epub 2021 Apr 8. German. PMID 33831971
- [Result] Dahmen A, Keller FM, Derksen C, Kotting L, Lippke S. [Which Digital Services do Psychosomatic Rehabilitation Patients Use During the Corona Pandemic and do Interrelations with Anxiety and Depressive Symptoms Exist?]. Psychother Psychosom Med Psychol. 2021 Dec;71(12):508-514. doi: 10.1055/a-1503-5548. Epub 2021 Sep 20. German. PMID 34544173
- [Result] Keller FM, Derksen C, Kotting L, Dahmen A, Lippke S. Distress, loneliness, and mental health during the COVID-19 pandemic: Test of the extension of the Evolutionary Theory of Loneliness. Appl Psychol Health Well Being. 2023 Feb;15(1):24-48. doi: 10.1111/aphw.12352. Epub 2022 Mar 9. PMID 35266309